CLINICAL TRIAL: NCT00077103
Title: Phase II Trial of Combined Modality Combretastatin A-4 Phosphate (CA4P)-Based Therapy for Patients With Newly Diagnosed Anaplastic Thyroid Cancer [Induction Chemotherapy With Doxorubicin/Cisplatin; Combined Modality Therapy With CA4P and Radiation; Followed by 2 Cycles of CA4P Consolidation]
Brief Title: Induction Chemotherapy Using Doxorubicin and Cisplatin Followed by Combretastatin A4 Phosphate and Radiation Therapy in Treating Patients With Newly Diagnosed Regionally Advanced Anaplastic Thyroid Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Panayiotis Savvides, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU3302; P30CA043703 (NIH); CASE-CWRU-3302 (Other: Case Comprehensive Cancer Center); CWRU-040337; OXIGENE-CWRU-3302
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Head and Neck Cancer
Keywords: anaplastic thyroid cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Thyroid Carcinoma, Anaplastic | interventions — Filgrastim; pegfilgrastim; Cisplatin; Doxorubicin; fosbretabulin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim — filgrastim (G-CSF) subcutaneously (SC) on days 3-21 or pegfilgrastim SC on day 2.
Biological: pegfilgrastim — filgrastim (G-CSF) subcutaneously (SC) on days 3-21 or pegfilgrastim SC on day 2.
Drug: cisplatin — cisplatin IV over 30-60 minutes on day 1
Drug: doxorubicin hydrochloride — doxorubicin IV over 5-10 minutes
Drug: fosbretabulin disodium — Combined Modality Phase:Patients also receive CA4P IV over 10 minutes weekly on the fifth day of radiotherapy. Beginning 4-6 weeks after the completion of the combined modality phase, patients receive CA4P IV over 10 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 2 courses.
  Other Names: Combretastatin A-4 Phosphate; CA4P
Radiation: radiation therapy — Beginning on day 22, patients undergo radiotherapy twice daily, 5 days a week, for 3-4 weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin and cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combretastatin A4 phosphate may stop the growth of cancer by stopping blood flow to the tumor. Combining doxorubicin and cisplatin with radiation therapy and combretastatin A4 phosphate may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving induction chemotherapy using doxorubicin and cisplatin together with radiation therapy and combretastatin A4 phosphate works in treating patients with newly diagnosed regionally advanced anaplastic thyroid cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in patients with newly diagnosed regionally advanced anaplastic thyroid cancer treated with induction chemotherapy comprising doxorubicin and cisplatin followed by combretastatin A4 phosphate (CA4P) and radiotherapy.
* Determine whether this regimen alters the natural history of anaplastic thyroid cancer by virtue of doubling the median survival of these patients from 10 to 20 months.

Secondary

* Determine a tolerable dose of CA4P when administered with radiotherapy in these patients. (Phase I portion of the study closed as of 5/6/04; patients now receive a fixed dose of CA4P)
* Determine the safety profile of this regimen in these patients.
* Determine clinical predictors of response (e.g., pretreatment tumor microvessel density and immature vessel staining, changes in sICAM-1 levels and tumor blood flow, and pharmacokinetic parameters) in patients treated with this regimen.
* Correlate the diminution in blood flow with tumor pain and response in patients treated with this regimen.

OUTLINE: This is a multicenter study of combretastatin A4 phosphate (CA4P). (Phase I portion of the study closed as of 5/6/04; patients now receive a fixed dose of CA4P)

* Induction phase: Patients receive doxorubicin IV over 5-10 minutes and cisplatin IV over 30-60 minutes on day 1. Patients also receive filgrastim (G-CSF) subcutaneously (SC) on days 3-21 or pegfilgrastim SC on day 2.
* Combined modality phase: Beginning on day 22, patients undergo radiotherapy twice daily, 5 days a week, for 3-4 weeks. Patients also receive CA4P IV over 10 minutes weekly on the fifth day of radiotherapy.

Cohorts of 6 patients receive 1 of 2 escalating doses of CA4P to determine a tolerable dose. The tolerable dose is defined as the dose at which less than 2 of 6 patients experience dose-limiting toxicity. (Phase I portion of the study closed as of 5/6/04; patients now receive a fixed dose of CA4P)

* Consolidation phase: Beginning 4-6 weeks after the completion of the combined modality phase, patients receive CA4P IV over 10 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 2 courses.

Treatment in all phases continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 1 year and then every 3 months for 2 years from study entry.

PROJECTED ACCRUAL: A total of 33 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed anaplastic or poorly differentiated variant thyroid carcinoma of either of the following:

  * Regionally advanced disease

    * Confined to the neck and/or superior mediastinum (i.e., above the level of the carina)
    * Measurable or evaluable* disease
  * Completely resected disease without measurable or evaluable disease NOTE: *At a minimum, abnormalities on physical exam or radiographic studies that may not be precisely measured but readily followed
* Must have original/diagnostic tumor blocks available to confirm histopathology and for tumor microvessel density immunohistochemistry

  * Patients with no available original/diagnostic tumor blocks must have tumor accessible for pretreatment needle core biopsy
* Must undergo indirect and direct laryngoscopy to ensure patency of the trachea/airway if deemed inoperable, with bulky thyroid/neck masses and/or suspicion of airway obstruction
* No distant metastases, including but not limited to, brain metastases, disease below the level of the carina, pulmonary parenchyma, and hepatic or bony metastases

  * Superior mediastinal disease (i.e., above the level of the carina) in addition to regional neck disease is allowed provided the disease can be contained in a single radiotherapy port

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 8.5 g/dL

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* ALT and AST ≤ 3.5 times upper limit of normal

Renal

* Creatinine ≤ 1.5 mg/dL

Cardiovascular

* LVEF ≥ 50% by echocardiogram
* EKG normal
* No prior angina
* No prior myocardial infarction (e.g., significant Q waves), QTc > 450 msec, or other clinically significant abnormalities on ECG
* No congestive heart failure
* No uncontrolled atrial arrhythmias or clinically significant arrhythmias, including any of the following:

  * Conduction abnormality
  * Nodal junctional arrhythmias and dysrhythmias
  * Sinus bradycardia or tachycardia
  * Supraventricular arrhythmias
  * Atrial fibrillation or flutter
  * Syncope or vasovagal episodes
* No significant heart wall abnormality or heart muscle damage by echocardiogram
* No uncontrolled hypertension (i.e., blood pressure consistently greater than 150/100 mm Hg irrespective of medication)

  * Hypertension is allowed provided there is clinical documentation of controlled blood pressure for 2 months before study entry
* No symptomatic peripheral vascular disease or cerebrovascular disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled hypokalemia or hypomagnesemia
* No concurrent serious infection
* No other nonmalignant uncontrolled medical illness or one whose control may be jeopardized by the complications of study therapy
* No grade 2 or greater pre-existing motor or sensory peripheral neuropathy
* No psychiatric disorder or other condition that would preclude study compliance
* No conditions associated with QTc prolongation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biologic therapy
* No concurrent immunotherapy

Chemotherapy

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy, except for the following:

  * Gonadotropin-releasing hormone agonists for patients with hormone-refractory prostate cancer
  * Hormone replacement therapy
  * Oral contraceptives
  * Megestrol for anorexia/cachexia

Radiotherapy

* No prior radiotherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* Prior attempt at resection or cytoreduction (e.g., debulking) surgery irrespective of surgical margins allowed provided there are no distant metastases
* At least 1 week but no more than 8 weeks since prior surgery and recovered

Other

* No other concurrent cytotoxic therapy
* No other concurrent antineoplastic therapy
* No other concurrent investigational therapy
* No concurrent medications known to prolong the QTc interval unless the medication can be held for at least 4 days during each treatment course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2003-11; Primary Completion 2007-02 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Median survival | at months 2, 4, 6, 8, 10, 12, 15, 18, 21, 24, 27, 30, 33, and 36

SECONDARY OUTCOMES:
Objective disease response | at the end of induction, combined modality therapy, and consolidation therapy, at 2 months after completion of consolidation therapy, at 2 month intervals during year 1, and then 3 month intervals during years 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Panayiotis Savvides, MD, Study Chair — Ireland Cancer Center at University Hosptials Case Medical Center, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Ireland Cancer Center at University Hosptials Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania